CLINICAL TRIAL: NCT04735692
Title: Impact of Periodontal Bacteria on the Effectiveness of Periodontal Therapy
Brief Title: Effectiveness of Periodontal Therapy on Periodontal Bacteria
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Catania (Other)
Responsible Party: Principal Investigator, Gaetano Isola, Researcher, University of Catania
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 02318
Record Dates: First submitted 2021-01-29; First posted 2021-02-03 (Actual); Last update posted 2022-12-16 (Actual); Status verified 2022-12

CONDITIONS: Periodontitis
MeSH Terms: conditions — Periodontitis

STUDY DESIGN:
Intervention Model Description: Patients undergo non-surgical quadrant scaling and root planing
Who Masked: Participant, Investigator
Masking Description: Both participants and clinicians were blinded to group and treatment assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Periodontitis quadrant Scaling root planing (Placebo Comparator): Patients undergo non surgical quadrant scaling and root planing performed per quadrant
  Interventions: Other: Full mouth or quadrant SRP
- Periodontitis full mouth scaling root planing (Active Comparator): Patients undergo non surgical full mouth scaling and root planing
  Interventions: Other: Full mouth or quadrant SRP

INTERVENTIONS:
Other: Full mouth or quadrant SRP — Full mouth or quadrant SRP

SUMMARY:
In light of the controversy that are already approved but that however still exists regarding the efficacy and influence of the protocols for the management of Periodontitis, the aim of this study was to evaluate, at 6 months follow-up, the post-treatment clinical parameters and immunological and gingival microbial profiles in patients with periodontitis, treated by either SRP in addition to full mouth scaling or quadrant scaling

DETAILED DESCRIPTION:
This trial was conducted in accordance with the World Medical Association's Declaration of Helsinki of 1975, and reviewed in 2008. The local ethical committee of the University of Messina approved the study protocol and each patient was carefully informed about the possible inherent risks of the study and provided their informed written consent 88 patients, aged 27 to 65 (mean age 57) were assessed for eligibility. In all subjects, subgingival plaque was acquired from 4 separate proximal sites at 180 days after therapy.

ELIGIBILITY:
Inclusion Criteria:

* Presence of at least 15 teeth
* CP with a minimum of 40% of sites with a clinical attachment level (CAL)

  ≥2mm and probing depth (PD) ≥4mm;
* Presence of at least ≥2 mm of crestal alveolar bone loss verified on digital periapical radiographs
* Presence of ≥40% sites with bleeding on probing (BOP)

Exclusion Criteria:

* Intake of contraceptives
* Intake of immunosuppressive or anti-inflammatory drugs throughout the last three months prior to the study
* Status of pregnancy or lactation
* Previous history of excessive drinking
* Allergy to local anaesthetic
* Intake of drugs that may potentially determine gingival hyperplasia such as Hydantoin, Nifedipine, Cyclosporin A or similar drugs.

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2021-02-05 (Actual); Primary Completion 2022-12-05 (Actual); Study Completion 2022-12-05 (Actual)

PRIMARY OUTCOMES:
Clinical attachment level | 1-year
  evaluation of changes in clinical attachment level

CONTACTS AND LOCATIONS:
Overall Officials: Gaetano Isola, Principal Investigator — Università degli Studi di Catania
Locations (1):
- University of Catania, Catania, CT, Italy

IPD SHARING:
Plan to Share IPD: Undecided
all collected IPD, all IPD that underlie results in a publication